CLINICAL TRIAL: NCT03500237
Title: Effectiveness of Internet-delivered Cognitive Behaviour Therapy for Chronic Conditions: Comparing Low Intensity Delivery Models
Brief Title: Internet-delivered Cognitive Behaviour Therapy for Chronic Conditions: Comparing Low Intensity Delivery Models
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Regina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-045
Record Dates: First submitted 2018-04-09; First posted 2018-04-18 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Anxiety; Depression; Chronic Disease
Keywords: anxiety; depression; internet-delivered cognitive behaviour therapy; randomized controlled trial; patient-centered; knowledge implementation; mental health system; therapist-assistance
MeSH Terms: conditions — Anxiety Disorders; Depression; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Team-Guided ICBT (Experimental): An 8-week transdiagnostic internet-delivered cognitive behavioural therapy (ICBT) for persons with chronic conditions course will be delivered to participants. In addition to the online program, a guide from the Online Therapy Unit team will provide support within one business day of the client's email. The team of guides consist of registered social workers, psychologists or supervised graduate students, with experience delivering ICBT. Amount of contact will be personalized to participants' needs.
  Interventions: Behavioral: Team-Guided ICBT
- Self-Guided ICBT (Active Comparator): An 8-week transdiagnostic internet-delivered cognitive behavioural therapy (ICBT) for persons with chronic conditions course will be delivered to participants. Participants are able to contact the Online Therapy Unit regarding any technical issues with logging onto the site. However, no psychological intervention will be provided. A team member from the Unit will contact the participant only if there is a significant clinical issue requiring attention (e.g., sudden increase in symptoms).
  Interventions: Behavioral: Self-Guided ICBT

INTERVENTIONS:
Behavioral: Team-Guided ICBT — An 8-week transdiagnostic internet-delivered cognitive behavioural therapy (ICBT) for persons with chronic conditions course will be delivered to participants. In addition to the online program, a guide from the Online Therapy Unit team will respond within one business day of the client's email. The team of guides consist of registered social workers, psychologists or supervised graduate students, with experience delivering ICBT. Amount of contact will be personalized to participants' needs.
  Arms: Team-Guided ICBT
Behavioral: Self-Guided ICBT — An 8-week transdiagnostic internet-delivered cognitive behavioural therapy (ICBT) for persons with chronic conditions course will be delivered to participants. Participants are able to contact the Online Therapy Unit regarding any technical issues with logging onto the site. However, no psychoeducational support will be provided. A team member from the Unit will contact the participant only if there is a significant clinical issue requiring attention (e.g., sudden increase in symptoms).
  Arms: Self-Guided ICBT

SUMMARY:
Chronic health conditions (e.g., heart disease, cancer, diabetes) represent any physical condition that persist for 3 months or more that requires ongoing management. Chronic health conditions are very common, and increase in prevalence with age. Internet-delivered Cognitive Behaviour Therapy (ICBT) is a promising approach for overcoming these barriers, and improving access to mental health care. In ICBT, clients receive content from traditional face-to-face CBT over the Internet, while receiving support and assistance from a guide through secure e-mail. The Chronic Conditions Course is an 8-week, 5 lesson ICBT program that consists of education and relapse prevention as well as cognitive, behavioural, and physical strategies for managing chronic conditions. This intervention has traditionally been delivered either with no support or with weekly brief (15 minute) individual therapist guidance via email and phone. However, in order to provide a faster response to clients using an on the demand (responding as quickly as possible and for sure within one business day team based approach (e.g., first available therapist responds) may be beneficial.

The proposed trial will examine the Chronic Conditions Course delivered by a team at the Online Therapy Unit based at the University of Regina versus a self-directed program. In the team based approach, participants will be able to contact the Online Therapy Unit if they have any questions regarding the content of the Chronic Conditions Course during the 8 week program. Participants in this group will receive a response from one of the members of the team within one business day. In the self-directed group, clients will receive automatic messages from the Online Therapy Unit that encourage participation during the 8 week program but otherwise will work on the course on their own. All participants will complete questionnaires prior to the start of the program, before each lesson of the program, once they have completed the program, and 3 months after completing the program. The primary outcome measures include anxiety and depression. Secondary outcomes include fatigue, pain, self-efficacy, disability, overall quality of life, and life satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* residing in Canada
* endorsing symptoms of anxiety or depression
* diagnosed with a chronic medical health condition
* chronic condition does not impact ability to complete treatment (ex. cognitive impairment)
* able to access a computer and internet service
* willing to provide a physician as emergency contact

Exclusion Criteria:

* high suicide risk
* suicide attempt or hospitalization in the last year
* primary problems with psychosis, alcohol or drug problems, mania
* currently receiving active psychological treatment for anxiety or depression
* not present in country during treatment
* concerns about online therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2021-08-24 (Actual); Study Completion 2021-08-24 (Actual)

PRIMARY OUTCOMES:
Change in depression | baseline, 8 weeks, 3 months
  Measured by Patient Health Questionnaire - 9 Item (PHQ-9)
Change in anxiety | baseline, 8 weeks, 3 months
  Measured by Generalize Anxiety Disorder - 7 Item (GAD7)

SECONDARY OUTCOMES:
Change in psychological distress | baseline, 8 weeks, 3 months
  Measured by Kessler 10-Item Scale
Change in disability | baseline, 8 weeks, 3 months
  Measured by World Health Organization Disability Assessment Schedule - 12 Item
Change in quality of life symptoms | baseline, 8 weeks, 3 months
  Measured by 5-level EuroQol-5D version (EQ-5D-5L), items are added for a score ranging from 5-25 with total score indicating: 5-14 Mild problem, 15-24 Moderate, 25 Worst Health State
Change in pain | baseline, 8 weeks, 3 months
  Measured by Brief Pain Inventory-Short Form
Change in fatigue | baseline, 8 weeks, 3 months
  Measured by Fatigue Symptom Inventory
Change in life satisfaction | baseline, 8 weeks, 3 months
  Measured by Satisfaction with Life Scale (SwLS), items are added together to get a score ranging from 5-35; Higher scores are indicative of greater life satisfaction
Change in self-efficacy | baseline, 8 weeks, 3 months
  Measured by Self-Efficacy for Managing Chronic Disease 6-item Scale
Change in treatment costs | baseline, 3 months
  Measured by Treatment Inventory of Costs in Psychiatric Patients (TIC-P) Adapted for Canada
Treatment credibility | baseline
  Measured by Treatment Credibility Questionnaire (TCQ) which contains 4 items. The first three items range from 0-9 with higher scores indicating better outcome, and the fourth item ranges from 0-100%, with higher scores indicating greater improvement in functioning.
Treatment satisfaction | 8 weeks
  Measured by Internet-CBT Treatment Satisfaction Measure

CONTACTS AND LOCATIONS:
Overall Officials: Heather Hadjistavropoulos, PhD, Principal Investigator — University of Regina
Locations (1):
- Online Therapy Unit, University of Regina, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mehta SH, Nugent M, Peynenburg V, Thiessen D, La Posta G, Titov N, Dear BF, Hadjistavropoulos HD. Internet-delivered cognitive behaviour therapy for chronic health conditions: self-guided versus team-guided. J Behav Med. 2022 Oct;45(5):674-689. doi: 10.1007/s10865-022-00346-x. Epub 2022 Aug 3. PMID 35921055